CLINICAL TRIAL: NCT02281266
Title: Investigator Initiated Study of Thymosin in HBV-related HCC
Brief Title: Thymalfasin Adjuvant Therapy in Hepatitis B Virus (HBV)-Related Hepatocellular Carcinoma (HCC) After Curative Resection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jia Fan (Other)
Collaborators: SciClone Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Jia Fan, Prof., Fudan University
Organization: Fudan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZDX-2014-05
Record Dates: First submitted 2014-10-15; First posted 2014-11-03 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: Curable Hepatitis B Virus-Related Hepatocellular Carcinoma
MeSH Terms: interventions — Thymalfasin; Nucleosides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- treatment (T) (Experimental): The patients of treatment arm will be administered subcutaneously Thymalfasin at dose of 1.6mg twice a week for 12 months after curative resection, followed by 12 months observation.
  Nucleoside analog plan to give to HBV DNA positive patients.
  Interventions: Procedure: curative resection; Drug: thymalfasin; Drug: nucleoside analog (suggest to use entecavir)
- control (C) (Other): The patients of control arm will be followed up for 2 years periodically after curative resection, without the investigational product (Thymalfasin) therapy.
  Nucleoside analog plan to give to HBV DNA positive patients.
  Interventions: Procedure: curative resection; Drug: nucleoside analog (suggest to use entecavir)

INTERVENTIONS:
Procedure: curative resection
Drug: thymalfasin — 1.6mg twice a week, 12 months
  Other Names: ZADAXIN
  Arms: treatment (T)
Drug: nucleoside analog (suggest to use entecavir)

SUMMARY:
Efficacy and safety of Thymalfasin adjuvant therapy in HBV-related HCC after curative resection.

DETAILED DESCRIPTION:
Multi-center, Randomized, Controlled Clinical Trial to Evaluate the Efficacy and Safety of Adjuvant Thymalfasin Therapy in Hepatitis B Virus (HBV)-Related Hepatocellular Carcinoma After Curative Resection.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria during perioperative period

* Male or female patients with age between 18-70 years.
* Life expectance ≥ 3 months.
* Diagnosis of Hepatocellular Carcinoma confirmed by Histological or Cytological examination.
* Hepatitis B history with current HBsAg positive and/or HBV DNA positive
* Will undergo hepatic curative resection.
* Tumor feature a. with cancer embolus b. a solitary nodule measuring between 3-8 cm or 2 nodule, a total combined measurement between 3-8 cm
* East Cooperative Oncology Group performance score of 0-2
* Normal liver function or sufficient liver function, defined as Chlid's-Pugh A

Inclusion criteria at baseline post-operation (4weeks ± 7days post-operation)

* No documented evidence of disease recurrence with computed tomography (CT) scan and CT angiography.
* Grade A of Chlid's-Pugh score
* hematological test white blood cell (WBC)>3.5X109/L, red blood cell (RBC)>30%, platelet count (PLT)>50,000/Ul, neutrophil (NEU)>1.0X109/L, Cr<1.5 mg/dl
* signed informed consent

Exclusion Criteria:

* Any anti-cancer therapy, including liver transplant, transarterial Chemo-embolization (TACE), image-guided tumor ablation, radiotherapy, chemotherapy, molecular targeted therapy and immunotherapy, etc. prior to the liver surgery procedure.
* Taking the hepatotoxic drug or immunosuppressant drug.
* Invasion of portal vascular and its first branch, hepatic duct and its first branch, inferior vena cava and hepatic vein.
* Organ transplant recipient.
* Extra-hepatic organs and lymph node metastasis.
* Uncontrolled Hypertension, unstable angina within 3 months, congestive heart failure (New York Heart Association (NYHA) Class II or greater), history of myocardial infarction within 6 months prior to randomization and severe arrhythmia need to be treated.
* History of malignancy other than a successfully treated non-metastatic cutaneous squamous cell or basal cell carcinoma and/or localized carcinoma in situ of the cervix
* Known human immune deficiency virus (HIV) infection
* hepatitis C virus (HCV) infection
* History of stroke or transient ischemic attack within 6 months prior to randomization
* Active or untreated central nervous system (CNS) metastasis
* History of clinically significant drug or alcohol abuse
* Prior treatment with immunomodulator (e.g. interferon, Thymalfasin) or traditional Chinese medicine within 30 days prior to randomization
* Know postoperative complications (e.g. infection, bleeding, bile leak) at baseline
* Known allergic reaction to the investigational product and its excipient.
* Female subjects who are pregnant or breast-feeding or considering becoming pregnant during the study.
* The investigator considers the subject, for any reason, to be unacceptable for study participation.
* Participating in other clinical trials of the drug or medical device within 30 days prior to randomization.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2015-01; Primary Completion 2018-06 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free Survival | 2-year

SECONDARY OUTCOMES:
Recurrence-free Survival (RFS) | 1-year
Overall survival (OS) | 1-year
Overall survival (OS) | 2-year
Mean recurrence time | up to 2 years
Tumor sample immune cell counts | tumor sample will be collected at baseline and when relapse
  immune cell counts includes T cell counts(CD3, CD4, CD8), Treg count(FoxP3), Th17 cell count(IL-17), natural killer(NK) cell count(CD56), neutrophil count(CD66b), Mφ count(CD68), dendritic cell(DC) count (CD1a,CD83), MVD(CD31)
incidence and types of Adverse Events (AE) and serious adverse event (SAE) | 2-year
  AE and SAE will be reported. The number of patients with AE and the number of patients with SAE will be calculated.
number of patients with abnormal laboratory value, vital signs and ECG result | 2-year
  The number of patients with abnormal laboratory value, vital signs and ECG result during the study will also be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Ge S, Huang D. Systemic therapies for hepatocellular carcinoma. Drug Discov Ther. 2015 Oct;9(5):352-62. doi: 10.5582/ddt.2015.01047. PMID 26632544
- [Derived] Qiu SJ, Zhou ZG, Shen F, Li AJ, Chen MS, Ying MG, Chen Z, Zhang YX, Sun HC, Fan J. A multicenter, randomized, observation-controlled clinical trial to evaluate the efficacy and safety of thymalfasin adjuvant therapy in patients with HBV-related HCC after curative resection - first announcement of the protocol. Expert Opin Biol Ther. 2015;15 Suppl 1:S133-7. doi: 10.1517/14712598.2015.1039979. Epub 2015 Jun 22. PMID 26094695